CLINICAL TRIAL: NCT05903118
Title: A Phase I/II, Randomized, Blind, Placebo-Controlled Study to Evaluate the Safety and Immunogenicity of SARS-CoV-2 mRNA Vaccine (RBMRNA-176) in Healthy Adults Aged 18 Years and Older
Brief Title: A Phase I/II Study to Evaluate a SARS-CoV-2 mRNA Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Argorna Pharmaceuticals Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CP-RBMRNA-001-02
Record Dates: First submitted 2023-06-12; First posted 2023-06-15 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: SARS-CoV-2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Participants aged 18 to 59 years. (Experimental): Escalating dose levels
  Interventions: Biological: RBMRNA-176
- Participants aged 60 years and older. (Experimental): Escalating dose levels
  Interventions: Biological: RBMRNA-176
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: RBMRNA-176 — Anti-viral RNA vaccine for active immunization against COVID-19 administered as intramuscular injection
  Arms: Participants aged 18 to 59 years.; Participants aged 60 years and older.
Other: Placebo — 0.9% sodium chloride (normal saline) injection
  Arms: Placebo

SUMMARY:
The phase I/II study is to evaluate the safety and immunogenicity of SARS-COV-2 mRNA Vaccine (RBMRNA-176) at different doses in healthy subjects aged 18 years and older.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years and older, Body Mass Index (BMI) is between 18-30, able to provide legal proof of identity
2. Participants voluntarily agreed to participate in the study and signed an informed consent form
3. The subject has ability to understand the research process and is willing and able to comply with all research proposals and other requirements of the study
4. Axillary temperature ≤37.3°C on the day of injection
5. Negative SARS-CoV-2 reverse transcription-polymerase chain reaction (RT-PCR) test, without infective history of severe acute respiratory syndrome (SARS), coronavirus disease 2019 (COVID-19), Middle East Respiratory Syndrome (MERS)
6. Female subjects of childbearing age are not at pregnant period (negative result of pregnancy test) or lactation period
7. Female subjects of childbearing age had taken effective contraceptive measures 1 month before enrollment
8. Female subjects of childbearing age and male subjects agree to use effective contraception for 12 months from the screening visit to the full injection
9. Female subjects of childbearing age and male subjects agree that do not donate eggs (eggs, oocytes) for assisted reproduction (female subjects of childbearing age) or avoid sperm donation (male subjects) from screening period until 12 months after injection

Exclusion Criteria:

1. Chest x - ray is clinically significant abnormal as determined by the investigators
2. The vital signs or examinations are clinically significant abnormal as determined by the investigators prior to randomization
3. A history of severe allergy (including drugs, vaccines, and foods) or to any component of the experimental vaccine, e.g., allergic shock, allergic laryngeal edema, anaphylactoid purpura, dyspnea, and angioedema, etc.
4. Subjects have been diagnosed with a serious disease, congenital malformation or chronic disease (including but not limited to: respiratory disease or chronic bronchitis such as asthma, serious cardiovascular disease, kidney disease, autoimmune disease, thrombocytopenic purpura, thalassemia, malignant tumor, hereditary allergic constitution, etc.) that may interfere with the conduct or completion of the study
5. Diagnosed with diseases may affect immune system function, congenital or acquired immune deficiency or suppression (e.g., tuberculosis, human immunodeficiency virus (HIV)), Hepatitis B, hepatitis C, syphilis infection, uncontrollable autoimmune disease, no spleen or spleen dysfunction
6. Lymph node - related diseases (such as lymphadenitis, lymph node adhesion, lymph node tuberculosis, tumor metastasis, etc.) or skin scars and fistulas at the lymph node site, or lymphadenopathy, tenderness, skin redness and swelling at the lymph node site within 7 days prior to injection
7. History or family history of convulsions, epilepsy, encephalopathy, psychiatry, or history of narcolepsy
8. Within 3 days prior to injection, an acute illness or attack of a chronic disease, or the use of antipyretic analgesic or anti - allergic drugs
9. Subjects have contraindications to intramuscular injection, such as having been diagnosed with thrombocytopenia, any blood clotting disorder or receiving anticoagulant therapy
10. Long-term use of immunopotentiator or immunosuppressant therapy within 6 months prior to the first dose injection (continuous orally or by injection for more than 14 days).
11. Use of any blood or blood - related products (e.g., blood transfusion, use of human albumin, human immunoglobulin, etc.) within 6 months prior to the first dose injection
12. Any blood lost > 400 mL within 28 days prior to the screening visit (e.g., donate blood or component blood, or injured), or plan to donate blood or component blood between the screening visit and 28 days after the last dose injection
13. Previously received any SARS-CoV-2 vaccine or plan to receive other SARS-CoV-2 vaccines
14. Other vaccines have been administered within 4 weeks prior to the first dose injection or other injection schedule (except for emergency injections such as Rabies vaccine and Tetanus vaccine) between the screening period and 28 days after the injection
15. Any abnormal or permanent body art (such as tattoos) at the site of the injection, which the researchers think to interfere with observing local reactions at the site of the injection
16. Female subjects planning to become pregnant or male subjects' partners planning to become pregnant from screening period to 12 months after whole schedule injection
17. Participating in or planning to participate in other clinical trials (drugs or vaccines) within 3 months prior to participating in this study
18. Other circumstances considered by the investigator as inappropriate to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2022-01-08 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-07-19 (Actual)

PRIMARY OUTCOMES:
Solicited local and systemic adverse reactions (AR) | Within 14 days after each dose
  For phase I
All Adverse Events (AE) related to injection | From the first dose to within 28 days after the whole schedule injection
  For phase I
The level of neutralizing antibody against SARS-CoV-2 | The 28th day after the whole schedule injection
  For phase II

SECONDARY OUTCOMES:
Unsolicited Adverse Events (AE) | After the first dose till before the second dose, and within 28 days after the second dose
  For phase I & II
All serious adverse events (SAE) | Within 21 days after the first dose, and within 28 days after the second dose, and 90days, 180 days, 360 days after the whole schedule injection
  For phase I & II
The level of Immunoglobulin G (IgG) antibody against SARS-CoV-2 S protein | The 21st day after the first dose, and the 7th day, 28th day, 90th day, 180th day, 360th day after the whole schedule injection
  For phase I & II
The level of neutralizing antibody against SARS-CoV-2 | The 21st day after the first dose, and the 7th day, 28th day, 90th day, 180th day, 360th day after the whole schedule injection
  For phase I
The level of neutralizing antibody against SARS-CoV-2 | The 21st day after the first dose, and the 7th day, 90th day, 180th day, 360th day after the whole schedule injection
  For phase II
Solicited local and systemic ARs | Within 14 days after each dose
  For phase II
All AEs related to injection | From the first dose to within 28 days after the whole schedule injection
  For phase II

CONTACTS AND LOCATIONS:
Locations (1):
- Chengdu Xinhua Hospital affiliated to North Sichuan Medical College, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No